CLINICAL TRIAL: NCT05012007
Title: Reminders for FIT (Fecal Immunochemical Test) Kits Via Different Modalities: a Randomized Controlled Trial
Brief Title: Reminder Modality for CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alaina Mori, Staff Physician, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: FIT2
Record Dates: First submitted 2021-06-22; First posted 2021-08-19 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer
Keywords: Cancer screening; Adherence
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm: No Reminder (No Intervention): Usual care
- Automated phone reminder (Experimental): Standard reminder via phone (audiocare)
  Interventions: Other: Reminder Phone
- Text reminder (Experimental): Standard reminder via text (VEText)
  Interventions: Other: Reminder Text

INTERVENTIONS:
Other: Reminder Phone — Standard reminder via phone (audiocare)
  Arms: Automated phone reminder
Other: Reminder Text — reminder via text (VEText)
  Arms: Text reminder

SUMMARY:
This is a randomized controlled trial that will evaluate the effectiveness of different reminder modalities for a population-based mailed FIT program at the VA Puget Sound among average risk Veterans who are due for annual colorectal cancer (CRC) screening.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial that will evaluate the effectiveness of two different reminder modalities in improving adherence to annual CRC screening.

Veterans eligible for enrollment into the trial will be randomized in a 1:1:1 allocation using permuted block randomization (with random block sizes of 3 and 6) to the following interventions:

1. Control arm: No reminder

   a. Intervention Type: No intervention
2. Arm 2: Automated phone reminder

   a. Intervention Type: Standard reminder via phone (audiocare)
3. Arm 3: Text reminder a. Intervention Type: Standard reminder via text (VEText)

Randomization will be stratified within arms by prior screening status (prior screener vs. never screener)

ELIGIBILITY:
Eligible participants are automatically enrolled in this project. We are unable to enroll participants upon request.

Inclusion Criteria:

* Veterans assigned to a primary care provider at the VA Puget Sound as of January 1, 2021
* At least 1 year of prior data available (evidence of at least one outpatient visit).
* Due for annual CRC screening

Exclusion Criteria:

* Not scheduled for either a screening or diagnostic colonoscopy within the following 12 weeks from assessment.
* No indication of current receipt of hospice care or record of recent death in the administrative data.
* No personal history of CRC or history of prior colectomy.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2653 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage of returned FIT Kits | three months post randomization
  the return rate at three months post randomization

SECONDARY OUTCOMES:
Percentage of returned FIT Kits | six months post randomization
  the return rate at six months post randomization

OTHER OUTCOMES:
Interim analysis | At 50% (n = 1327) of estimated sample size
  z-statistic will be calculated from the proportional difference between the combined treatment groups (all reminders) vs. control

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, MD, Principal Investigator — VA Puget Sound Health Care System; Stefanie Deeds, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deeds S, Schuttner L, Wheat C, Gunnink E, Geyer J, Beste L, Chen A, Dominitz JA, Nelson K, Reddy A. Automated Reminders Enhance Mailed Fecal Immunochemical Test Completion Among Veterans: a Randomized Controlled Trial. J Gen Intern Med. 2024 Jan;39(1):113-119. doi: 10.1007/s11606-023-08409-8. Epub 2023 Sep 20. PMID 37731137